CLINICAL TRIAL: NCT03227705
Title: Canadian Study on the Association of Pessary With Progesterone
Acronym: CAPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Centre hospitalier de l'Université de Montréal (CHUM) (Other); CHU de Quebec-Universite Laval (Other); St. Justine's Hospital (Other); Jewish General Hospital (Other); The Ottawa Hospital (Other); Queen's University (Other)
Responsible Party: Principal Investigator, Jean-Charles Pasquier, MD, PhD, MD, PhD, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13-159
Record Dates: First submitted 2017-07-12; First posted 2017-07-24 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Preterm Birth; Short Cervix
Keywords: Preterm birth; Short cervix; Pessary; Progesterone
MeSH Terms: conditions — Premature Birth | interventions — Progesterone; Pessaries

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravaginal progesterone (Active Comparator): Once the participant agrees and signs the consent form, the use of prophylactic progesterone will begin (PROMETRIUM, 200 mg in total of progesterone, 2 vaginal capsules per day at bedtime up to 36 6/7 weeks of gestation, Merck Canada Inc.)
  Interventions: Drug: Prometrium
- Intravaginal progesterone and pessary (Experimental): Once the participant agrees and signs the consent form, the use of prophylactic progesterone will begin (PROMETRIUM, 200 mg in total of progesterone, 2 vaginal capsules per day at bedtime, Merck Canada Inc.). Also, a perforated pessary (Dr. Arabin, cerclage pessary perforated) will be inserted. The pessary will be removed and the progesterone treatment will be stopped at 36 6/7 weeks of gestation.
  Interventions: Drug: Prometrium; Device: Dr. Arabin, cerclage pessary perforated

INTERVENTIONS:
Drug: Prometrium — Intravaginal use, off label, of Prometrium
  Other Names: Progesterone
Device: Dr. Arabin, cerclage pessary perforated — A Dr. Arabin, cerclage pessary perforated will be inserted participants diagnosed with a short cervix
  Other Names: Pessary
  Arms: Intravaginal progesterone and pessary

SUMMARY:
Prematurity is the leading cause of neonatal morbidity causing more than 1 million deaths worldwide per year. In 2012, a randomized controlled trial (RCT) testing "pessary" (silicone ring placed around the cervix) versus "no pessary" in patients with a short cervix showed a 4-fold reduction in the rate of spontaneous prematurity <34 weeks of gestation and a reduction in perinatal morbidity and mortality. This result was not found in a subsequent RCT and another study on the subject had to be stopped in the face of slow recruitment. Currently, the obstetric scientific community believes that other RCTs are needed before using the pessary in the clinic as a therapeutic option to prevent prematurity in the presence of a short cervix. However, before starting a large RCT, it is important to test the feasibility of recruitment.

DETAILED DESCRIPTION:
Hypothesis: A standardized recruitment process could allow the inclusion of 0.9% patient (CI 95%: 0,78-1.04) among women receiving a 18-23 weeks ultrasound scan.

Recruitment: Participants will be recruited, in a three-step manner, among women appointing for the 18-23 weeks ultrasound scan; i) assessment of the cervical length by abdominal ultrasound, ii) an endovaginal ultrasound measurement will be performed if the cervical length is ≤ 30 mm, iii) enrollment and consent of the patient to the pilot study, under the confirmation of the presence of a short cervix (≤ 25 mm) by the endovaginal ultrasound.

Intervention: Vaginal progesterone (200 mg/day, PROMETRIUM®, Merck Canada Inc.) until 37 weeks. Perforated cerclage pessaries (Dr. Arabin GmbH & Co. KG) will be placed in specialized clinic and will be removed at 37 weeks.

Size of the sampling and statistical analysis: This multicenter pilot study will be conducted in High-Risk Pregnancies Clinics in Quebec and in Ontario.

Over the 12 months period, the investigators expect to collect data from 26 000 abdominal ultrasounds. In accordance with the anticipated recruitment level of 0.9%, the investigators planned on enrolling 250 women. Within those women, 125 will be assigned randomly to the "progesterone" group and 125 to the "progesterone and pessary" group (1:1 ratio).

Perspective: This pilot study is designed to identify the challenges and provide strategies to deal with them in a larger study. Providing its feasibility, this study will lead to a definitive randomized controlled trial (including over 70 centers) to test the effectiveness of pessary and progesterone in preventing preterm birth.

ELIGIBILITY:
Inclusion Criteria:

* patient with a short cervix equal to or less than 25 mm by transvaginal ultrasound
* gestational age between 18 (0/7) and 23 (6/7) weeks of gestation according to the results of the ultrasound of the first trimester, or by integrating the date of the last period
* patients who were informed of the study and agreed to sign the consent form.

Exclusion Criteria:

* pregnancy with a fetus with a major congenital malformation - regular and painful uterine activity - history of preterm premature rupture of membranes (PPROM) - active vaginal bleeding - complete and incomplete placenta previa - cerclage of the cervix in place - antecedent of conisation - multiple gestation - ballooning of membranes outside the cervix into the vagina - allergy/intolerance or hypersensitivity to progesterone or any of its ingredients - chronic medical conditions that would interfere with study participation or evaluation of treatment - vaginal administration of another drug.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Recruitment feasibility | Up to 24 weeks (18 to 42 weeks of gestation)
  According to the anticipated recruitment rate, 0.9% of women having an anatomy scan could be included (95% CI, 0.78- 1.04). We will determine the % of women included in the study (until the 42 week of gestation) over women that received a anatomy scan.

SECONDARY OUTCOMES:
Preterm delivery | Before 34 weeks
  The secondary outcome is to determine the occurrence of spontaneous preterm births before 34 weeks in the progesterone alone group " without pessary harm ".

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Pasquier, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (8):
- Canada (8):
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Hospital, Ottawa, Ontario
  - Centre hospitalier de l'Université de Montréal, Montreal, Quebec
  - CHU Sainte-Justine, Montreal, Quebec
  - CIUSSS du Centre Ouest-de-l'Île-de Montréal, Montreal, Quebec
  - St.Mary's Hospital Center, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdel-Aleem H, Shaaban OM, Abdel-Aleem MA, Aboelfadle Mohamed A. Cervical pessary for preventing preterm birth in singleton pregnancies. Cochrane Database Syst Rev. 2022 Dec 1;12(12):CD014508. doi: 10.1002/14651858.CD014508. PMID 36453699